CLINICAL TRIAL: NCT00554502
Title: Supportive Versus Immunosuppressive Therapy for the Treatment Of Progressive IgA Nephropathy
Acronym: STOP-IgAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Verena Deserno, Clinical Trials Centre Aachen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP-IgAN
Record Dates: First submitted 2007-10-29; First posted 2007-11-07 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Palliative Care; Immunosuppression Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: supportive therapy with: ACE-inhibitor / ARB / Statin
- B (Active Comparator)
  Interventions: Drug: supportive and immunosuppressive therapy

INTERVENTIONS:
Drug: supportive therapy with: ACE-inhibitor / ARB / Statin — * Antihypertensive therapy with a target blood pressure below 125/75 mmHg (following current clinical guidelines).
  * ACE-inhibitors (ARB when an ACE-inhibitor is not tolerated)
  * Other antihypertensive medications depending on the clinical decision and following current guidelines.
  * Statin therapy
  * Dietary counseling for a low-sodium diet and, if GFR is below 60 ml/min, for a protein intake of 0.8 g/kg/day.
  Arms: A
Drug: supportive and immunosuppressive therapy — * supportive therapy as outlined above
  * depending on GFR:
    * methylprednisolone and prednisolone
    * cyclophosphamide and prednisolone; after 3 months azathioprine with prednisolone
  * Concomitant medication with the immunosuppressive treatment following current clinical practice
  Arms: B

SUMMARY:
* Evaluation of the efficacy of an immunosuppressive therapy added to a comprehensive supportive therapy to induce a clinical remission in patients at risk for progressive IgAN
* Investigation of differences between the treatments regarding the number of patients loosing more than 15 ml/min of GFR.

DETAILED DESCRIPTION:
The best treatment of glomerular diseases of the kidney is currently not well defined. This study aims to answer if in patients with IgA nephropathy, the most common type of glomerulonephritis an immunosuppressive treatment (with the use of steroids and chemotherapy) added to a supportive treatment is more effective than a supportive treatment alone (with the use of drugs lowering the blood pressure and the urinary protein loss).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients from 18-70 years with histologically proven primary IgAN with typical mesangioproliferative features. Diagnosis has to be made by a neuropathologist.
* Proteinuria above 0.75 g/day within 12 weeks prior to or at the first visit in the run-in phase (month -6)and presence of at least one further risk factor for the development of end stage renal disease

  1. arterial hypertension, defined as ambulatory blood pressure >140/90 mm Hg or the use of antihypertensive medication or
  2. impaired renal function, defined as creatinine clearance or estimated GFR <90 ml/min.

Exclusion Criteria:

* Known allergy or intolerance to study medication (except in case of ACE-inhibitor, in which case a change to an angiotensin receptor blocker is possible).
* Women who are pregnant or breastfeeding and women without sufficient contraception.
* Any prior immunosuppressive therapy.
* Variants of primary IgAN (e.g. rapidly progressive IgAN with crescents in >50% of glomeruli or minimal change GN with glomerular IgA deposits).
* Significant liver dysfunction (more than three fold increased GPT compared to norm)
* Contraindication for immunosuppressive therapy, like

  * acute or chronic infectious disease incl. hepatitis and HIV positive patients
  * any malignancy
  * leukocytopenia, thrombocytopenia or known allergy against prednisolone, cyclophosphamide or azathioprine
  * active intestinal bleeding, active gastric or duodenal ulcer
  * Need of permanent immunosuppression, (e.g. transplanted patients, steroid-dependent inflammatory diseases)
* Secondary IgAN or diseases associated with glomerular deposits of IgA.
* Additional other chronic renal disease.
* Creatinine clearance below 30 ml/min (mean of 3 measurements).
* Alcohol or drug abuse
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* Participation in a parallel clinical trial or participation in another clinical trial within the last 3 months.
* Subjects who are in any state of dependency to the sponsor or the investigators.
* Employees of the sponsor or the investigators.
* Subjects who have been committed to an institution by legal or regulatory order.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2008-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Patients reaching full clinical remission of their disease | at the end of the 3 year study period.
GFR loss of 15 ml/min or higher from baseline GFR | at the end of the 3 year study period

SECONDARY OUTCOMES:
-Absolute GFR-change. | at the end of the 3 years study period
GFR loss >=30 ml/min from baseline GFR | at the end of the 3 year study period
-Onset of end stage renal disease. | at the end of the 3 years study period
Mean annual change in one over serum creatinine concentration | at the end of the 3 years study period
Proteinuria at 12 and 36 months | 12 and 36 months
Disappearance of microhematuria | at the end of the 3 years study period

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Floege, Prof. Dr., Principal Investigator — Medical Clinic II, University Hospital Aachen
Locations (34):
- Germany (34):
  - Medical Clinic II, University Hospital Aachen, Aachen
  - 2. Medizinische Klinik, Nephrologie, Klinikum Augsburg, Augsburg
  - Campus Charité Mitte, Medizinische Klinik - Schwerpunkt Nephrologie, Centrum 13, Berlin
  - Charité Campus Virchow-Klinikum, Medizinische Klinik / Nephrologie, Berlin
  - Helios-Klinikum Berlin-Buch, Nephrologie Charité CCB, Berlin
  - St. Joseph Krankenhaus Medizinische Klinik II, Berlin
  - Klinikum Bremen-Mitte, Medizinische Klinik III, Bremen
  - Uniklinik Köln, Klinik IV für Innere Medizin, Nephrologie und Allgemeine Innere Medizin, Cologne
  - Universitätsklinikum Dresden, Medizinische Klinik III, Bereich Nephrologie, Dresden
  - Universitätsklinikum Düsseldorf, Klinik für Nephrologie, Düsseldorf
  - Universitätsklinikum Erlangen, Medizinische Klinik IV, Erlangen
  - Universitätsklinikum Essen, Klinik für Nieren- und Hochdruckkrankheiten, Essen
  - Universitätsklinikum Freiburg, Innere Medizin IV, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg GmbH, Medizinische Klinik und Poliklinik II, Giessen
  - Universitätsklinikum Göttingen, Zentrum Innere Medizin, Abteilung für Nephrologie und Rheumatologie, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, 3. Medizinische Klinik und Poliklinik, Hamburg
  - Medizinische Hochschule Hannover, Abteilung Nephrologie, Hanover
  - Med. Universitätsklinik Heidelberg, Nierenzentrum Heidelberg, Sektion Nephrologie, Heidelberg
  - Universitätsklinikum Jena, Medizinische Klinik III, Jena
  - Westpfalz-Klinikum GmbH, Abteilung für Nephrologie und Transplantationsmedizin, Kaiserslautern
  - Universitätsklinikum Magdeburg, Klinik für Nephrologie, Zentrum für Innere Medizin, Magdeburg
  - Dialysezentrum am Brand, Mainz
  - Universitätsklinikum Mannheim, V. Medizinische Klinik, Mannheim
  - Universitätsklinikum Marburg, Klinik für Innere Medizin, Schwerpunkt Nephrologie, Marburg
  - KfH Nierenzentrum, München
  - Klinikum der LMU, Nephrologisches Zentrum, München
  - Klinikum rechts der Isar, Medizinische Klinik II, Abteilung für Nephrologie, München
  - Universitätsklinikum Münster, Medizinische Klinik und Poliklinik D, Münster
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Innere Medizin II, Regensburg
  - Krankenhaus der Barmherzigen Brüder, Abteilung Innere Medizin II, Trier
  - Universitätsklinikum Tübingen, Medizinische Klinik IV, Sektion für Nieren- und Hochdruckkrankheiten, Tübingen
  - Dialyse-Zentrum Dres.med. PD H. Reichel, Th. Weinreich u. C., Villingen-Schwenningen
  - Zentrum für Nieren- und Hochdruckkrankheiten, Wiesbaden
  - Universitätsklinik Würzburg, Medizinische Klinik und Poliklinik I, Würzburg

REFERENCES:
- [Derived] Alladin A, Hahn D, Hodson EM, Ravani P, Pfister K, Quinn RR, Samuel SM. Immunosuppressive therapy for IgA nephropathy in children. Cochrane Database Syst Rev. 2024 Jun 12;6(6):CD015060. doi: 10.1002/14651858.CD015060.pub2. PMID 38864363
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Rauen T, Eitner F, Fitzner C, Sommerer C, Zeier M, Otte B, Panzer U, Peters H, Benck U, Mertens PR, Kuhlmann U, Witzke O, Gross O, Vielhauer V, Mann JF, Hilgers RD, Floege J; STOP-IgAN Investigators. Intensive Supportive Care plus Immunosuppression in IgA Nephropathy. N Engl J Med. 2015 Dec 3;373(23):2225-36. doi: 10.1056/NEJMoa1415463. PMID 26630142
- [Derived] Yeo SC, Liew A, Barratt J. Emerging therapies in immunoglobulin A nephropathy. Nephrology (Carlton). 2015 Nov;20(11):788-800. doi: 10.1111/nep.12527. PMID 26032537
- [Derived] Eitner F, Ackermann D, Hilgers RD, Floege J. Supportive Versus Immunosuppressive Therapy of Progressive IgA nephropathy (STOP) IgAN trial: rationale and study protocol. J Nephrol. 2008 May-Jun;21(3):284-9. PMID 18587715